CLINICAL TRIAL: NCT03582904
Title: Using tDCS to Enhance Learning of a New Walking Pattern
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Pilot data suggested the paradigm would need significant revision.
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Susanne M Morton, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1240484
Record Dates: First submitted 2018-06-14; First posted 2018-07-11 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: no Condition Being Studied; tDCS Only in Healthy Subjects
Keywords: motor learning; tDCS; locomotion
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS (Experimental): Anodal transcranial direct current stimulation (tDCS) targeting the primary motor cortex delivered via saline-soaked sponge electrodes (anode, 8 cm^2; cathode 38.4 cm^2) at an intensity of 1.5 milliamperes over < 30 minutes.
  Interventions: Procedure: tDCS
- Control (Sham Comparator): Anodal transcranial direct current stimulation (tDCS) targeting the primary motor cortex delivered via saline-soaked sponge electrodes (anode, 8 cm^2; cathode 38.4 cm^2) at an intensity of 1.5 milliamperes over 2 minutes.
  Interventions: Procedure: tDCS

INTERVENTIONS:
Procedure: tDCS — real or sham tDCS delivered to primary motor cortex

SUMMARY:
The ability to change walking patterns is important for daily tasks such as stepping over an obstacle. This change of walking pattern can occur in a strategic manner, i.e., consciously making one step longer or shorter. Healthy individuals can learn a new walking pattern through perturbed visual feedback of their walking information (Kim et al., 2015; Kim et al., 2017). This type of learning is thought to largely involve explicit strategy. Transcranial direct current stimulation (tDCS) is a form of non-invasive brain stimulation that can enhance learning of some motor tasks (Reis et al., 2009), and primarily has been studied in the upper extremity. In locomotor learning, prior recent work by the investigators has suggested that tDCS does not affect non-strategy based locomotor learning, and the investigators speculate that tDCS may benefit learning of strategic tasks instead. The purpose of this study is to determine if tDCS can enhance learning and retention of a new walking pattern in a strategy-based, visually guided locomotor task in healthy individuals. Two groups of young, healthy participants will be recruited to learn a new walking pattern through perturbed visual feedback, with retention of learning tested on the second day. One group will receive tDCS, which is expected to enhance learning. The other group will receive placebo stimulation and serve as a control. Results from this work will provide information on which type of motor learning is sensitive to enhancement with tDCS, and may help pave the path for utilizing tDCS for neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Medically stable and generally healthy
* Able to walk on a treadmill without the use of handrails for 20 minutes at a speed of 1.0 m/s without rest
* Resting heart rate ≤100 beats per minute
* Resting blood pressure ≤140/90 mm Hg
* Willing and able to attend all testing sessions

Exclusion Criteria:

* Any chronic or recent medical conditions, including any musculoskeletal, cardiovascular, pulmonary, psychiatric or neurological diagnosis
* Any impaired sensation or weakness in either lower extremity
* History of serious traumatic head injury, defined as a loss of consciousness for more than 5 minutes and/or requiring medical treatment
* Any history of acute or chronic problems with balance or more than 1 fall in the last 12 months
* History of brain surgery
* Taking 4 or more medications
* Current or chronic pain located anywhere in the body
* History of seizures
* Currently pregnant (if a female of childbearing age)
* Currently taking any medications that act on the central nervous system
* Implanted pumps or stimulators above the shoulders
* Metal aneurysm, other metal surgical clip placement, or any other metal in the head, face, or neck, except for dental fillings

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Magnitude of Locomotor Learning | study day 1
  Step length produced on the perturbed leg at the end of the learning period on study day 1 and subtracted from baseline (pre-learning period) step length
Magnitude of Locomotor Learning Retention | study day 2
  Step length produced on the perturbed leg on study day 2, normalized to the Magnitude of Locomotor Learning achieved on study day 1

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Morton, PhD, PT, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No